CLINICAL TRIAL: NCT05778006
Title: Multi-Center Registry for ME/CFS, Including ME/CFS Following Epstein-Barr Virus-Associated Infectious Mononucleosis (EBV-IM) or Coronavirus Disease 2019 (Covid-19)
Brief Title: Multi-Center Registry for ME/CFS
Acronym: MECFS-R
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: MECFS-R
Record Dates: First submitted 2023-03-20; First posted 2023-03-21 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: ME/CFS; CFS/ME; ME/CFS Following EBV-associated Infectious Mononucleosis; ME/CFS Following COVID-19
Keywords: ME/CFS; CFS/ME; SARS-CoV-2; COVID-10; Post-COVID-19 condition; Chronic fatigue syndrome; Myalgic encephalomyelitis; Epstein-Barr virus; EBV
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: None Retained — Serum samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ME/CFS study (MECFS-R) aims to create a large-scale registry that provides data on epidemiology, phenotypes, and disease trajectories of and health care for ME/CFS at any age in Germany, which can be used for future clinical trials.

DETAILED DESCRIPTION:
ME/CFS (ICD-10 G93.3) is a multisystem chronic disease that can lead to severe disability. Pre-pandemic prevalence was estimated at approximately 0.3% worldwide, and increasing prevalence is observed due to ME/CFS in the context of long-term sequelae of coronavirus diseases 2019 (COVID-19). In Germany, the number of affected people in Germany was estimated as approximately 350.000-400.000 in 2018/2019 and almost 500.000 in 2021. ME/CFS can manifest at any age, with peak prevalence in adolescents and young adults. Common triggers include COVID, influenza, and Epstein-Barr virus-associated infectious mononucleosis (EBV-IM). Non-infectious triggers are known as well. Autoimmunity and dysfunction of the autonomic nervous system (ANS) were suggested as possible pathomechanisms. Core symptoms include fatigue, post-exertional malaise (PEM), and unrefreshing sleep. Additional symptoms comprise cognitive deficits ("brain fog"), orthostatic intolerance, neuroendocrine, and immunological symptoms. ME/CFS is diagnosed according to clinical criteria (mostly criteria by the Institute of Medicine (IOM) or Canadian Consensus Criteria) and by appropriate differential diagnostics to exclude other disorders with similar symptoms. So far, no biomarker or specific therapy is available. Therapeutic approaches are holistic and aim at the palliation of symptoms as well as psychosocial support. Self-management with pacing is recommended. Knowledge of ME/CFS among healthcare providers is still scarce, and many patients do not receive adequate care.

With this web-based, German-wide registry, the investigators aim at deep phenotyping of the disease, identification of subtypes and risk factors, describing trajectories of the disease and patient journeys, and providing clinical data for future clinical trials. Patients are also invited to contribute biosamples for future translational research.

ELIGIBILITY:
Inclusion Criteria:

* ME/CFS diagnosis (ICD-10 G93.3) based on internationally established criteria
* Informed consent by patients and/or guardian(s)

Exclusion Criteria:

* No ME/CFS (ICD-10 G93.3)
* No informed consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ME/CFS
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2052-05-31 (Estimated); Study Completion 2052-05-31 (Estimated)

PRIMARY OUTCOMES:
Phenotyping ME/CFS: Medical History | 30 years
  Routine assessment of the medical history, such as current and previous medication, vaccinations, comorbidities, and more, to achieve a profound ME/CFS phenotype.
Assessment of routine physical examination findings | 30 years
  Routine physical examination to achieve a profound and detailed ME/CFS phenotype.
Number of participants with abnormal laboratory tests results | 30 years
  Measurement of a routine set of laboratory parameters including blood tests (cell count[cell/µl], C-reactive protein [mg/dl], immunoglobulins A/M/G [md/dl], antinuclear antibodies [titer], etc.) and urine/stool analysis (e.g. calprotectin [mg/kg], positive hemoglobin in urine test stripe) to achieve a profound ME/CFS phenotype.
Number of participants with abnormal technical exam results | 30 years
  Technical exams (e.g. restrictive and obstructive pattern in pulmonary function tests, conduction in electrocardiography, ultrasound imaging, magnetic resonance imaging, etc.) will be performed as indicated to achieve a profound and detailed ME/CFS phenotype.

SECONDARY OUTCOMES:
Evaluation of Patient Journeys | 30 years
  Patients' journeys will be analyzed regarding the specialization of involved physicians visited, time to diagnosis, and time to treatment.
Definition of Sub-cohorts | 30 years
  Using routine data, sub-cohorts will be identified.
Prevalence of Comorbidities | 30 years
  Prevalence of comorbidities of patients with ME/CFS will be analyzed.
Identification of Candidate Prognostic Markers | 30 years
  Correlation of routine clinical data (e.g., medical history, routine laboratory, and physical examination) with clinical outcome (e.g., health-related quality of life, disease severity, and social participation).

CONTACTS AND LOCATIONS:
Overall Officials: Uta Behrends, Prof. Dr. med., Principal Investigator — MRI Chronic Fatigue Center for Young People (MCFC) Children's Hospital, Technical University of Munich & Munich Municipal Hospital
Locations (1):
- MRI Chronic Fatigue Center for Young People (MCFC) Children's Hospital, Technical University of Munich & Munich Municipal Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hieber H, Pricoco R, Gerrer K, Heindrich C, Wiehler K, Mihatsch LL, Haegele M, Schindler D, Donath Q, Christa C, Grabbe A, Kircher A, Leone A, Mueller Y, Zietemann H, Freitag H, Sotzny F, Warlitz C, Stojanov S, Hattesohl DBR, Hausruckinger A, Mittelstrass K, Scheibenbogen C, Behrends U. The German Multicenter Registry for ME/CFS (MECFS-R). J Clin Med. 2024 May 28;13(11):3168. doi: 10.3390/jcm13113168. PMID 38892879